CLINICAL TRIAL: NCT05932186
Title: Interscalene Block Versus Upper Trunk Block in Shoulder Arthroscopy: Randomized Comparative Study of the Ease Between the Two Techniques Among Residents
Brief Title: Upper Trunk Block Feasibility by Anesthesia Residents
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0306047
Record Dates: First submitted 2023-04-28; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-04

CONDITIONS: Anesthesia, Local; Shoulder Pain
Keywords: Anesthesia, Local; Shoulder
MeSH Terms: conditions — Shoulder Pain | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interscalene block (Active Comparator): Patients will receive inter scalene brachial plexus block combined with general anesthesia
  Interventions: Procedure: Interscalene brachial plexus block combined with general anesthesia
- Upper trunk block (Active Comparator): Patients will receive upper trunk brachial plexus block combined with general anesthesia
  Interventions: Procedure: Upper trunk brachial plexus block combined with general anesthesia

INTERVENTIONS:
Procedure: Interscalene brachial plexus block combined with general anesthesia — Baseline diaphragmatic assessment will be performed before the nerve block in the sitting position. Interscalene block will be done as follows. US probe will be placed slightly lower to the level of the cricoid cartilage, followed by scanning of the neck to search for C5 and C6 nerve roots enclosed between the anterior and middle scalene muscles. The needle will be introduced in-plane from lateral to medial through the middle scalene muscle until the tip enters the brachial plexus sheath between the C5 and C6 roots, where LA will be injected.
  Patients will be transported to the operation room where general anaesthesia will be induced with tracheal intubation Fentanyl (0.5 μg/kg) will be given to maintain the heart rate and mean blood pressure 20% lower than preinduction values. Intravenous 1 gram paracetamol and 8 mg dexamethasone will be given to all patients as part of multimodal analgesia
  Arms: Interscalene block
Procedure: Upper trunk brachial plexus block combined with general anesthesia — Baseline diaphragmatic assessment will be performed before the nerve block in the sitting position like the the ISB group
  Upper trunk will be visualized distal to the convergence of the C5 and C6 nerve roots but proximal to the departure of the suprascapular nerve (This nerve is a small hypoechoic circle that depart the lateral aspect of the upper trunk and courses posterolateral under the omohyoid muscle). The needle will be introduced in-plane from lateral to medial under the deep cervical fascia and through a very small portion of the middle scalene muscle, until the needle tip lies adjacent to the upper trunk, LA will be distributed below and above the upper trunk. Scanning for the upper trunk can be started from the supraclavicular fossa and moving proximal or opposite to cricoid cartilage and moving distal.
  The following steps will be done as in the ISB group
  Arms: Upper trunk block

SUMMARY:
The study compares between the success rate of interscalene block and upper trunk block performed by anesthesia trainee for intra and postoperative analgesia during shoulder arthroscopy. The duration of performing the block, guidance intervention by the consultant and block failure will be recorded.

DETAILED DESCRIPTION:
Investigators hypothesize that upper trunk block (UTB) is not inferior to interscalene brachial plexus block (ISB) regarding analgesia, easier to perform, with superior success rates, and less side effects in shoulder arthroscopy surgeries when undertaken by anaesthesia trainee.

A sample of 120 patients {60 patients in ISB group and 60 patients in UTB group} is needed to detect difference in 20% in rate of success of block also this sample is sufficient to detect difference in {Duration of the block performance, visualization of the anatomic structures and Consultant guidance, with a power 80% at a significance level of 05. Sample size was calculated using Number Cruncher Statistical Systems (NCSS) 2004 and Process Automation Software System (PASS) 2000 program Patients will be excluded if they have severe pulmonary disease, allergy to any of the study medications, local infection at any of the puncture sites, chronic gabapentin or pregabalin use, chronic opioid use, preexisting neuropathy of the operative limb, herniated cervical disc, or body mass index more than 35 kg/m2.

Upon arrival to the block room, the procedure will be explained to patients and a written informed consent will be obtained. Patients will be randomly categorized into two equal groups (group ISB and group UTB) using a numbered sealed envelope method. All blocks will be performed guided by a 5-13 MHz linear ultrasound (US) probe of a Sonosite (M-Turbo; Sonosite Inc, Bothell, W, USA) portable US machine.

Baseline diaphragmatic assessment will be performed before the nerve block in the sitting position. A curved array 3-5 MHz transducer of a Sonosite (M-Turbo; Sonosite Inc, Bothell, W, USA) portable US machine will be placed inferior to the costal margin in a longitudinal orientation at the anterior axillary line on the left or in the midclavicular line on the right. The ultrasound beam will be directed medially and cephalad to visualize the posterior third of the hemi-diaphragm by using either the spleen or the liver as an acoustic window, relatively. First the view will be obtained in a two-dimensional B-mode then the M-mode sonography will be used to quantify the extent of diaphragmatic excursion between full inspiration and full expiration once a view of the curved, hyperechoic diaphragmatic line has been obtained. This assessment will be carried out by the research anaesthetist.

Blocks will be carried out by anaesthesia residents who have one year experience in ultrasound guided regional anesthesia under direct supervision of a consultant anaesthetist (After demonstrating five successive blocks in each technique). Patients, surgeons, and the research anaesthetist will be blinded to the block technique.

All patients will be attached to a multichannel monitor and a venous catheter will be inserted in the dorsum of the hand of the unoperated limb. Intravenous sedation with 2 mg midazolam will be given. After tilting the extended neck to the contralateral side while the patient in the supine position, all blocks will be preceded by local anaesthetic infiltration (2-3 mL of lidocaine 1%) after applying the Standard disinfection. The local anaesthetic (LA) mixture that will be used (10 ml bupivacaine 0.25 %) in both groups.

Nerve blocks:

Group ISB:

The US probe will be placed slightly lower to the level of the cricoid cartilage, followed by scanning of the neck to search for C5 and C6 nerve roots enclosed between the anterior and middle scalene muscles. The needle will be introduced in-plane from lateral to medial through the middle scalene muscle (preferably in the upper third of the muscle to avoid injuring the dorsal scapular and long thoracic nerves) until the tip enters the brachial plexus sheath between the C5 and C6 roots, where LA will be injected. Back tracing from the supraclavicular fossa could be done instead to reach the interscalene groove.

Group UTB:

The upper trunk will be visualized distal to the convergence of the C5 and C6 nerve roots but proximal to the departure of the suprascapular nerve (This nerve is a small hypoechoic circle that depart the lateral aspect of the upper trunk and courses posterolateral under the omohyoid muscle). The needle will be introduced in-plane from lateral to medial under the deep cervical fascia and through a very small portion of the middle scalene muscle, until the needle tip lies adjacent to the upper trunk, LA will be distributed below and above the upper trunk. Scanning for the upper trunk can be started from the supraclavicular fossa and moving proximal or opposite to cricoid cartilage and moving distal.

An additional of 5 mL of the same LA mixture will be injected after performing each block superficial to the middle scalene muscle and prevertebral fascia, to block the supraclavicular nerves (lower branches of the superficial cervical plexus having C3-4 nerve roots, supplying the ''cape'' area of the shoulder) in both groups.

The duration of performing the block by the residents will be recorded, which is the time between the beginning of US scanning and needle withdrawal from the patients' neck. Inability to perform the block by residents either due to inability to specify the nerve structure correctly or to follow the needle tip during injection will be guided by the consultant and will be recorded as a guidance intervention. Guidance interventions are verbal instructions that guide the resident either to modify the image of the anatomic structures of interest by probe manipulations or to modify the needle tip path in a certain direction. Any block that will take more than 10 minutes to be performed or taken over by the consultant, will be considered a failure. Successful block performance (primary aim) is the completion of the block within 10 minutes with or without verbal guidance from the consultant.

After block performance, sensory and motor blockade will be assessed every 5min for 30min. Motor block will be evaluated by asking the patient to abduct his arm and will be graded on a three-points scale (2 = normal; 1 = weakness, and 0 = complete loss of power). Sensory block will be evaluated in the C4, C5, and C6 dermatomes and will be graded on a three-points scale (2 = normal; 1 = loss of sensation to pinprick; and 0 = loss of sensation to light touch). Block success will be defined as a sensory score of 0 within 30min.

Thirty minutes after block performance in the block room diaphragmatic excursion will be reassessed by the same research anaesthetist who did the baseline assessment before the block, as he is blinded to the block given. Complete hemi-diaphragmatic paralysis will be defined as a 75 to 100% decrease in excursion compared to baseline or the occurrence of paradoxical movement. Partial and absent hemi-diaphragmatic paresis will be defined as 25 to 75% decrease or a less than 25% decrease in diaphragmatic excursion, respectively.

Patients will be transported to the operation room where general anaesthesia will be induced with tracheal intubation using intravenous propofol (1.5 to 2.0 mg/kg), rocuronium (0.6 to 0.8 mg/kg), and fentanyl (1 μg/kg). Anaesthesia will be maintained with isoflurane/air-oxygen mixture. An additional fentanyl (0.5 μg/kg) will be given to maintain the heart rate and mean blood pressure 20% lower than preinduction values. Intravenous 1 gm paracetamol and 8 mg dexamethasone will be given to all patients as part of multimodal analgesia.

After surgery, all patients will be transferred to the post-anaesthesia care unit (PACU) until meeting the discharge criteria. Pain at rest will be measured using an 11-point numerical rating visual analogue scale (VAS), intravenous 6 mg of nalbuphine will be given if VAS ≥4 and total nalbuphine consumption will be recorded during the postoperative hospital stay. Once oral intake is tolerated, all patients will receive multimodal analgesia consisting of oral paracetamol 1 gm every 8 hours and oral celecoxib 200mg every 12 hours.

ELIGIBILITY:
Inclusion Criteria

* Patients aged 18 to 75 years
* American Society of Anesthesiologists physical status I to III
* Scheduled for arthroscopic rotator cuff repair Exclusion criteria
* Severe pulmonary disease
* Allergy to any of the study medications
* Local infection at any of the puncture sites
* Chronic gabapentin or pregabalin use
* Chronic opioid use
* Preexisting neuropathy of the operative limb, herniated cervical disc
* Body mass index more than 35 kg/m2.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-07-15 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Success rate of upper trunk block and interscalene block | 30 minutes after block performance
  Sensory and motor blockade will be assessed 30 minutes after block performance. Motor block will be evaluated by asking the patient to abduct his arm and will be graded on a three-points scale (2 = normal; 1 = weakness, and 0 = complete loss of power). Sensory block will be evaluated in the C4, C5, and C6 dermatomes and will be graded on a three-points scale (2 = normal; 1 = loss of sensation to pinprick; and 0 = loss of sensation to light touch). Block success will be defined as a sensory score of 0 within 30min

SECONDARY OUTCOMES:
Duration of performing the block | During the procedure
  Time between the beginning of US scanning and needle withdrawal from the patients' neck
Guidance interventions | During the procedure
  (Number of Verbal instructions that guide the resident either to modify the image of the anatomic structures of interest by probe manipulations or to modify the needle tip path in a certain direction)
Visualization of anatomic structures | During the procedure
  5 point scale [5-point scale according to the block given. Either the C5-6 roots or upper trunk (anterior division, posterior division, and suprascapular nerve), Very good = clearly recognizable as monofascicular or bifascicular, Good = perfectly identifiable, but presence of fascicles not clearly recognizable, Acceptable = blurry nerve structures, but good contrast between nerve roots and adjacent muscles, Poor = blurry nerve roots and muscles, Very poor = identification of nerve roots and muscles not possible]
Postoperative pain | 24 hours postoperatively
  Pain at rest will be measured using an 11-point numerical rating visual analogue scale (VAS). 10 is the worst pain ever and 0 is no pain
Opioid consumption | 24 hours postoperatively
  Intravenous 6 mg of nalbuphine will be given if VAS ≥4 and total nalbuphine consumption will be recorded during the postoperative hospital stay
Complications | 24 hours postoperatively
  Number

CONTACTS AND LOCATIONS:
Overall Officials: Moustafa A Moustafa, MD, Principal Investigator — Alexandria University, Faculty of Medicine
Locations (1):
- Alexandria Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Upon request
Supporting Information: Study Protocol, SAP
Time Frame: One year
Access Criteria: Email of principal investigator

REFERENCES:
- [Result] Abdallah FW, Halpern SH, Aoyama K, Brull R. Will the Real Benefits of Single-Shot Interscalene Block Please Stand Up? A Systematic Review and Meta-Analysis. Anesth Analg. 2015 May;120(5):1114-1129. doi: 10.1213/ANE.0000000000000688. PMID 25822923